CLINICAL TRIAL: NCT02246985
Title: Bioavailability of Carotenoids Incorporated Into Processed Foods: Bread and Mayonnaise
Brief Title: Bioavailability of Carotenoids Added Into Processed Foods
Acronym: CAROTFoods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 14/HSMC/2010
Record Dates: First submitted 2014-09-18; First posted 2014-09-23 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2016-03

CONDITIONS: Cardiovascular Disease
Keywords: Processed foods; Carotenoids in plasma, urine and faeces; alpha-carotene; beta-carotene; Vitamin A; Lycopene; Gut absorption; Bread; Mayonnaise; Bioavailability; Fruits and Vegetables; Inflammation; Oxidative Stress
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Plain bread with plain mayonnaise (Experimental): Control meal. The bread and mayonnaise in this meal does not have vegetable powders incorporated into them, hence this meal does not contain carotenoids
  Interventions: Dietary Supplement: Control
- Vegetable bread only (Experimental): A vegetable powder (carrot and tomato) containing bread portion will be served alone. The amount of vegetable powder in the bread will be standardised to contain a known amount of carotenoids
  Interventions: Dietary Supplement: Vegetable bread only
- Vegetable bread with plain mayonnaise (Experimental): A vegetable powder (carrot and tomato) containing bread portion will be served with plain mayonnaise. The amount of vegetable powder in the bread will be standardised to contain a known amount of carotenoids.
  Interventions: Dietary Supplement: Vegetable bread with plain mayonnaise
- Plain bread with vegetable mayonnaise (Experimental): Plain bread will be served with a vegetable powder (carrot and tomato) containing mayonnaise. The amount of vegetable powder in the mayonnaise will be standardised to contain a known amount of carotenoids.
  Interventions: Dietary Supplement: Plain bread with vegetable mayonnaise

INTERVENTIONS:
Dietary Supplement: Control — The bread and mayonnaise in this meal does not have vegetable powders incorporated into them. Hence this meal does not contain carotenoids.
  Other Names: plain bread with plain mayonnaise
  Arms: Plain bread with plain mayonnaise
Dietary Supplement: Vegetable bread only — A vegetable powder (carrot and tomato) containing bread portion will be served alone. The amount of vegetable powder in the bread portion will be standardised to contain a known amount of carotenoids.
  Arms: Vegetable bread only
Dietary Supplement: Plain bread with vegetable mayonnaise — Plain bread will be served with a vegetable powder (carrot and tomato) containing mayonnaise. The amount of vegetable powder in the mayonnaise will be standardised to contain a known amount of carotenoids.
  Arms: Plain bread with vegetable mayonnaise
Dietary Supplement: Vegetable bread with plain mayonnaise — A vegetable powder (Carrot and tomato) containing bread portion will be served with plain mayonnaise. The amount of vegetable powder in the bread portion will be standardised to contain a known amount of carotenoids
  Arms: Vegetable bread with plain mayonnaise

SUMMARY:
Carotenoids are a family of pigments found abundantly in fruits and vegetables. They are responsible for the colour of many fruits and vegetables such as tomatoes, melon, peppers and orange coloured fruits and vegetables. Carotenoids such as beta-carotene are important for the human body as precursors of vitamin A. They are also thought to be important as anti-oxidants and may help protect against cancer and heart disease. Although many foods are rich sources of carotenoids poor bioavailability often limits the amounts that are absorbed and available for metabolism in humans.

Devising practical ways and means of increasing carotenoid bioavailability could lead to better health outcomes. Processed foods are now widely eaten by many, both for their taste and convenience. No studies have thus far looked at the bioavailability of carotenoids that have been added into processed foods. Thus the purpose of this study is to investigate the bioavailability of carotenoids that have been incorporated into processed food products (bread and mayonnaise).

DETAILED DESCRIPTION:
Carotenoids are a diverse group of natural-occurring fat-soluble pigments. Whilst over 600 different types have been characterised around 20 have been found in human tissue in the postprandial state, however, over 90% of these absorbed carotenoids are made up of 6 specific types (alpha-Carotene, beta-carotene, Lycopene, Lutein, Zeaxanthin and Cryptoxanthin)

There is good evidence to suggest that carotenoids play a notable role in human health both through their pro-vitamin activity and as biological antioxidants. Carotenoids are believed to be responsible for the beneficial effects of fruits and vegetables in preventing human chronic diseases such as cancer and cardiovascular disease. Increasing fruit and vegetables intakes in individuals can sometimes be difficult and unsustainable, therefore, increasing bioavailability may be an effective alternative approach to maximise health outcomes.

A notable number of vegetables are rich sources of carotenoids, however, the amounts available to the human body for metabolism are often small due to poor bioavailability. For instance, studies have shown that bioavailability of carotenoids from carrots and tomatoes can be as low as 1-3%. The bioavailability of carotenoids has been shown to depend on factors such as their source, degree of cooking, processing, mechanical breakdown, presence of fat and interactions between carotenoids. Whilst the presence of fat significantly increases carotenoid absorption, the oil type, quantity and form it is in all affect bioavailability.

Recent work suggests that carotenoid bioavailability improves when fat is present in the form of mayonnaise rather than as plain oil. This may be due to the emulsion properties of mayonnaise which allows better solubilisation of amphiphilic compounds such as carotenoids. Mayonnaise has also been shown to be more miscible in gastric juices (compared to plain oil) and this too may be contributing to the greater absorption of carotenoids.

The present study builds upon this previous work and studies carotenoid bioavailability in processed food systems. Using a bread-mayonnaise meal the study compares carotenoid bioavailability when it is incorporated either into the bread or the mayonnaise. Furthermore, the study investigates the impact of mayonnaise on the bioavailability of carotenoids incorporated into a processed food (bread). The study will focus on the bioavailability of three principle carotenoids found in foods, alpha-carotene, beta-carotene and lycopene. Carrot and tomato are used as the sources of carotenoids.

HYPOTHESIS Carotenoid bioavailability is influenced by the food matrix in which they are contained.

OBJECTIVES

1. To compare the acute-phase bioavailability (systemic and gut absorption) of targeted carotenoids (alpha-carotene, beta-carotene and lycopene) when they are incorporated into the different processed food matrices (bread and mayonnaise)
2. Study how mayonnaise affects the acute bioavailability of carotenoids incorporated into a processed food.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females Aged between 18 and 75 years. Body mass index between 18.5 - 40 kg/m2. Blood pressure equal to or less than 139/89 mmHG. HbA1C less than or equal to 6.5%. Total blood cholesterol less than 6.0mmol/l

Exclusion Criteria:

* Suffering from Diabetes, kidney disease, hepatic disease, gout, gastrointestinal disorder, thromboembolic or coagulation disease, hypertension, thyroid disorder or hypercholesterolaemia On prescription medications Orlistat, Digoxin, Anti-arrhythmics, tricyclic anti-depressants, neuroleptics, oral anti-diabetic medication, insulin, anti-inflammatories, anti-pyretics and Statins Allergic/Intolerant to any of the foods in the study Vegetarian or Vegan Restricted eating and/or eating disorders Alcohol and/or substance abuse Regularly take nutritional supplements (once a day) Smoking Poor venous access and veins difficult to cannulate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-03 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in Carotenoid concentrations in plasma and in chylomicron-rich fraction | At baseline, at every hour for up to 8 hours postprandial and at 24hours after test meal
  Carotenoids in plasma and in the chylomicron-rich fraction will be measured using reverse-phase HPLC

SECONDARY OUTCOMES:
Change in carotenoid concentration in urine | at baseline and at every hour for up to 8 hours post-prandial and at 24hours after test meal
  Carotenoids in urine will be measured using reverse-phase HPLC

OTHER OUTCOMES:
Measurement of plasma retinol and retinyl ester concentrations | at baseline and at every hour for up to 8 hours post-prandial and at 24 hours after the test meal
  Plasma retinol and retinyl ester concentrations will be measured using reverse-phase HPLC
Plasma cholesterol concentrations | At baseline and at every hour for up to 8 hours post-prandial and at 24hours after the test meal
  Plasma cholesterol concentrations will be measured using reverse-phase HPLC
Satiety and palatability of test meals | immediately before and after consumption of test meals
  Measured using 100mm continuous-line visual analogue scales anchored at each end with opposing answers to satiety and palatability related questions

CONTACTS AND LOCATIONS:
Overall Officials: Viren Ranawana, Msc, PhD, Principal Investigator — Rowett Institute of Nutrition & Health, University of Aberdeen, Greenburn Road, Bucksburn, Aberdeen,, United Kingdom AB21 9SB
Locations (1):
- Rowett Institute of Nutrition and Health, Human Nutrition Unit, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No